CLINICAL TRIAL: NCT01895842
Title: Phase I Study of Ruxolitinib for Patients With Low or Intermediate-1 Risk Myelodysplastic Syndrome (MDS)
Brief Title: Ruxolitinib for Patients With Low or Intermediate-1 Risk Myelodysplastic Syndrome (MDS)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013-0012; NCI-2013-02204 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2013-07-05; First posted 2013-07-11 (Estimated); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Leukemia
Keywords: Leukemia; Myelodysplastic syndrome; MDS; Low or intermediate-1 risk; Maximum tolerated dose; MTD; Ruxolitinib; Jakafi; INCB018424; INC424
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes | interventions — ruxolitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ruxolitinib (Experimental): Part 1: Dose of ruxolitinib received will depend when patient joined study. The first group of patients receive the lowest dose of ruxolitinib. Starting dose level for Part 1, 5 mg by mouth twice a day for a 28 day cycle. The second group of patients receive the lowest dose of ruxolitinib for 1 cycle and if no intolerable side effects are seen, the dose will increase to the next higher dose for Cycles 2 and beyond. The third group of patients receive the higher dose taken by the second group for 1 cycle and if no intolerable side effects are seen, the dose will be increased for Cycles 2 and beyond. The fourth group of patients take the higher dose taken by the third group for 1 cycle and if no intolerable side effects are seen, the dose will increase to the next higher dose for Cycles 2 and beyond.
  If patients enrolled in Part 2, they will receive ruxolitinib at the highest dose that was tolerated in Part 1.
  Interventions: Drug: Ruxolitinib

INTERVENTIONS:
Drug: Ruxolitinib — Starting dose level for Part 1: 5 mg by mouth twice a day for a 28 day cycle.
  Starting dose level for Part 2: Maximum tolerated dose from Part 1.
  Other Names: Jakafi; INCB018424; INC424

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of ruxolitinib that can be given to patients with low or intermediate-1 risk MDS. The safety of this drug will also be studied, and whether it can help to control the disease.

DETAILED DESCRIPTION:
Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to a study group based on when you join this study. Up to 4 groups of 3-6 participants will be enrolled in Part 1 of the study, and up to 7 participants will be enrolled in Part 2.

If you are enrolled in Part 1, the dose of ruxolitinib you receive will depend on when you joined this study. The first group of participants will receive the lowest dose of ruxolitinib. The second group of participants will receive the lowest dose of ruxolitinib for 1 cycle and if no intolerable side effects are seen, the dose will increase to the next higher dose for Cycles 2 and beyond. The third group of participants will receive the higher dose taken by the second group for 1 cycle and if no intolerable side effects are seen, the dose will be increased for Cycles 2 and beyond. The fourth group of participants will take the higher dose taken by the third group for 1 cycle and if no intolerable side effects are seen, the dose will increase to the next higher dose for Cycles 2 and beyond.

If you are enrolled in Part 2, you will receive ruxolitinib at the highest dose that was tolerated in Part 1.

Study Drug Administration:

Each cycle is 28 days.

You will take ruxolitinib by mouth 2 times a day (about 12 hours apart), with or without food.

Study Visits:

One (1) time a week during Cycles 1 and 2 and then on Day 1 of Cycles 3 and beyond, blood (about 2-3 teaspoons) will be drawn for routine tests. On Day 28 of each cycle and Day 1 of Cycles 3 and beyond, this blood may also be used for cytogenetic testing if your doctor thinks it is needed.

On Day 28 of Cycles 1 and 2 and then every 3 cycles, you will have a bone marrow aspiration to check the status of the disease and for cytogenetic testing, if your doctor thinks it is needed.

On Day 28 of Cycle 1 and Day 1 of Cycles 3 and beyond, you will have a physical exam.

If the doctor thinks it is needed, urine will be collected on Day 1 of each cycle for routine tests.

Length of Dosing:

You may continue taking the study drug for up to 2 years. You will no longer be able to take the study drug if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on the study will be over after the end-of-dosing visit.

End-of-Dosing Visit:

After you are finished taking the study drug:

* You will have a physical exam.
* You will have a bone marrow aspiration to check the status of the disease.
* Blood (about 2-3 teaspoons) will be drawn for routine tests. This blood may also be used for cytogenetic testing if your doctor thinks it is needed.

Follow-up Visit:

About 30 days after the End-of-Dosing visit, a member of the study team will contact you by phone. You will be asked how you are feeling and about any side effects you may be experiencing. This phone call should take 10-15 minutes.

This is an investigational study. Ruxolitinib is FDA approved and commercially available for the treatment of myelofibrosis. Its use in this study is investigational. The study doctor can explain how ruxolitinib is designed to work.

Up to 31 participants will be enrolled in this study. All will take part at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with previously treated low or intermediate-1 risk MDS by the IPSS classification (this is defined in table 1)
2. Patients must have one of the following: elevated b2-microglobulin levels (defined as 2 times compared to normal), carry a JAK2 mutation, or presence of phosphorylated p65 NF-kB component in at least 5% of bone marrow cells.
3. Signed informed consent indicating that patients are aware of the investigational nature of this study in keeping with the policies of UTMDACC.
4. Age >/= 18 years old
5. Prior therapy with growth factor support, lenalidomide, 5-azacytidine, decitabine or other investigational agents are allowed. A four week wash out period will be required before receiving study medication.
6. Patients must have the following non-hematologic values Aspartate aminotransferase (AST/SGOT) and alanine aminotransferase (ALT/SGPT) </= 2.5 x Upper Limit of Normal (ULN) or </= 5.0 x ULN if hepatic involvement is present; Serum bilirubin </= 2 x ULN; Serum creatinine </= 2 x ULN or 24-hour creatinine clearance >/= 60 ml/min
7. Patients with Childbearing potential must agree to use appropriate forms of birth control

Exclusion Criteria:

1. Previously untreated low or intermediate-1 risk MDS patients because there are approved therapies for these patients.
2. Uncontrolled undercurrent illness that in the opinion of the treating physician would contraindicate the use of the drug.
3. Patients with active infections including uncontrolled HIV infection, active hepatitis B, C, or any other symptomatic systemic infection requiring active therapy will be excluded from study
4. Patients receiving potent CYP3A4 (such as but not limited to boceprevir, clarithromycin, conivaptan, grapefruit juice, indinavir, itraconazole, ketoconazole, lopinavir/ritonavir, mibefradil, nefazodone, nelfinavir, posaconazole, ritonavir, saquinavir, telaprevir, telithromycin, voriconazole) inhibitors will be excluded from the study.
5. Women who are pregnant or lactating.
6. Patients with a white blood cell count of more than 30x10^3 K/uL will not be eligible for this study.
7. Patients that have received prior allogeneic stem cell transplantation are excluded from this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2014-02 (Actual); Primary Completion 2019-04-02 (Actual); Study Completion 2019-04-02 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Ruxolitinib | 28 days
  Maximum tolerated dose (MTD) is the maximum dose at which <33% of patients experience a dose limiting toxicity (DLT). Dose limiting toxicity defined as any grade 3 or higher non-hematologic toxicity.

SECONDARY OUTCOMES:
Number of Participants with Response of Ruxolitinib | 8 weeks
  Criteria for response follows the modified International Working Group (IWG) response criteria for altering natural history of MDS defined as: Complete Remission, Partial Remission, Stable Disease, Cytogenetic Response, Disease Progression.

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Garcia-Manero, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Abaza Y, Hidalgo-Lopez JE, Verstovsek S, Jabbour E, Ravandi F, Borthakur G, Estrov Z, Alvarado Y, Burger J, Schneider H, Soltysiak KA, Wei Y, Kantarjian HM, Bueso-Ramos CE, Garcia-Manero G. Phase I study of ruxolitinib in previously treated patients with low or intermediate-1 risk myelodysplastic syndrome with evidence of NF-kB activation. Leuk Res. 2018 Oct;73:78-85. doi: 10.1016/j.leukres.2018.09.004. Epub 2018 Sep 14. PMID 30245189
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org